CLINICAL TRIAL: NCT06958978
Title: Effects of QUANTUM Probe for Skin Rejuvenation and Subdermal Retraction in Patients Undergoing High-Definition Liposculpture
Acronym: Quantum001
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Total Definer Research Group (Other)
Responsible Party: Principal Investigator, Alfredo Hoyos, Plastic Surgeon, Total Definer Research Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Quantum
Record Dates: First submitted 2025-02-02; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Skin Laxity; Skin Tightening; Body Contouring Surgery; Skin Elasticity; Skin Firmness; Liposuction
Keywords: Quantum; Quantum RF; Elastometer; Body contouring; Liposuction; Liposculpture; High Definition Liposculpture
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: All patients will receive Quantum Radiofrequency device as intervention in the anatomical areas were the skin laxity requires treatment. The skin laxity variables will be collected for all the areas at baseline (after liposculpture), immediate after Quantum, and during follow up months 1, 3, and 6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Quantum RF (Experimental): Right after the Liposuction procedure is completed, introduce the Quantum RF probe through the incision ports used for the liposuction. Using an imaginary grid with 1x1 cm pattern, apply assuring even distribution the Quantum RF (energy 15 J, pulse mode 3.0 pps) in the anatomical area. Maintain a uniform pace and energy level across the grid, covering both superficial and deep layers, to avoid hotspots and ensure consistent results.
  Interventions: Device: Quantum RF

INTERVENTIONS:
Device: Quantum RF — Patented handpiece device designed for skin rejuvenation and tightening through intraoperative subdermal Radiofrequency treatment.

SUMMARY:
This prospective study aims to evaluate the safety and effectiveness of Quantum, a fully internal bipolar radiofrequency probe, for the treatment of prominent skin laxity, providing patients with a more toned and youthful appearance, in patients undergoing High-Definition (HD) Liposculpture.

The main questions this study seeks to answer are:

* Does Quantum reduce skin laxity in patients undergoing HD Liposculpture?
* Is the effectiveness in skin laxity reduction influenced by demographical factors, including age, gender, and phototype?

The participants will be adult patients (between 18-60 years) undergoing HD Liposculpture, with any measurable degree of skin laxity. The participants can not be pregnant, have history of scaring/healing problems, autoimmune diseases, severe dermatological conditions, have metal implants, be obese, or have important comorbidities.

DETAILED DESCRIPTION:
Study design: Interventional prospective cohort study, non-randomized, non-controlled, no masking.

Eligible patients will be approached, the study aims, objectives, procedures, and voluntary participation will be explained. In case patient consent to participate, a written informed consent will be signed. The patients will be comprehensively evaluated by the plastic surgeon, and the areas selected for Quantum use, will be chosen according to the degree of skin laxity of the anatomical region.

Data Collection:

* Demographic, Clinical, and surgical variables are going to be collected in an Excel-based password protected database.
* Other procedure related variables are also going to be collected in the same database, hemoglobin and hematocrit levels, time to discharge, and complications.
* The effect of the intervention in the skin laxity will be measured with Elastometer after liposculpture before Quantum, right after Quantum use, 1, 3 and 6 months post procedure. Variables to collect will include area, skin thickness, elasticity, viscoelasticity, and time to retraction.
* Satisfaction Scores: Global Aesthetic Improvement Scale (GAIS) evaluated at least 3 months postoperatively.
* Photographical records will be kept with images pre procedure, and at follow up 1, 3, and 6 months.

The study procedures include:

* Procedure: All patients will undergo the standardized HD Liposculpture technique. Measurements of skin laxity will be performed with the Elastometer. Using the same ports of Liposculpture, Quantum device will be inserted, and the radiofrequency energy used in recommended parameters (energy 15 J, pulse mode 3.0 pps). Once the procedure is finished, with the patient still in operating table take the first post-treatment skin laxity measurements.
* Post procedure follow up: Skin laxity measurements with Elastometer in 1, 3, and 6 months postoperative controls.

Study Locations: Dhara Clinic (Bogota, Colombia)

Ethical Considerations:

* IRB Approval: The study will adhere to the Declaration of Helsinki principles and will be approved by an Institutional Review Board (IRB).
* Informed Consent: Participants will be provided comprehensive information about study procedures, risks, and benefits, and written consent will be obtained.
* Data Confidentiality: All participant data will be anonymized and securely stored.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing body contouring procedures (liposuction or liposculpture), either individually or combined with a maximum of two other major aesthetic procedures involving face, breast, or dermolipectomy.
* Healthy patients without underlying comorbidities (classified as ASA≤II)

Exclusion Criteria:

* Pregnant patients, patients planning to get pregnant, or in breastfeeding stage
* Past medical history of any collagen disease or autoimmune conditions, including lupus, scleroderma, connective tissue disorders, rheumatoid arthritis, or multiple sclerosis.
* Past medical history of skin disease including active skin infections, dermatitis, or history of keloid formation.
* Patient with any metal implants or pacemakers
* BMI ≥ 32 kg/m2.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Skin elasticity | 6 months
  Objectively calculate using Elastometer the difference in the skin elasticity measures pre Quantum use (but after liposculpture procedure), immediate after Quantum use, and in the postoperative follow up on the 1st, 3rd and 6th month.
Skin Viscoelasticity | 6 months
  Objectively calculate using Elastometer the difference in the skin viscoelasticity measures pre Quantum use (but after liposculpture procedure), immediate after Quantum use, and in the postoperative follow up on 1st, 3rd and 6th month
Skin retraction time | 6 months
  Objectively calculate using Elastometer the difference in the retraction time measures pre Quantum use (but after liposculpture procedure), immediate after Quantum use, and in the postoperative follow up on 1st, 3rd and 6th month

SECONDARY OUTCOMES:
Patient satisfaction | 6 months
  Patient-reported satisfaction scores measured using Global Aesthetic Improvement Scale (GAIS) for the reduction of skin laxity, and improvement of the appearance.
  The GAIS is a standardized scale used primarily in cosmetic and dermatological treatments to assess the overall aesthetic improvement of a patient after a procedure. It consist of three questions:
  * how do you feel about your appearance after surgery? Possible answers: Very much improved, much improved, slightly improved, no change.
  * Are you satisfied with the surgery? Very satisfied, satisfied, not satisfied.
  * Would you recommend the surgical procedure? Possible answers: Yes, perhaps, no.

CONTACTS AND LOCATIONS:
Locations (1):
- Dhara clinic, Bogotá, DC, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Depending upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: After results publication in scientific manuscript
Access Criteria: Request to the main author, stating the aims of the request, and the use the data will be given

REFERENCES:
- [Background] Ibrahiem SMS. Aesthetic Nonexcisional Arm Contouring. Aesthet Surg J. 2022 Jun 20;42(7):NP463-NP473. doi: 10.1093/asj/sjac031. PMID 35170726
- [Background] Chia CT, Theodorou SJ, Hoyos AE, Pitman GH. Radiofrequency-Assisted Liposuction Compared with Aggressive Superficial, Subdermal Liposuction of the Arms: A Bilateral Quantitative Comparison. Plast Reconstr Surg Glob Open. 2015 Aug 10;3(7):e459. doi: 10.1097/GOX.0000000000000429. eCollection 2015 Jul. PMID 26301148
- [Background] Cala Uribe LC, Perez Pachon ME, Babaitis R, Zannin Ferrero A, Aljure Diaz MF. Variable Energy and Ultrasound-based Liposculpture of the Arms: Multicenter and Multidevice Study. Plast Reconstr Surg Glob Open. 2024 Mar 19;12(3):e5649. doi: 10.1097/GOX.0000000000005649. eCollection 2024 Mar. PMID 38948160